CLINICAL TRIAL: NCT04352686
Title: Effects of Serotonin Agonist Buspirone on Multimodal Esophageal Stimulation in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Busprione MuMoS HV
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone (Active Comparator): Buspirone 20 mg per oral
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Administration of buspirone to assess esophageal sensitivity
  Arms: Buspirone
Drug: Placebo — Administration of placebo to assess differences in esophageal sensitivity
  Arms: Placebo

SUMMARY:
To investigate if buspirone, a partial 5-HT-1A receptor agonist, is able to modify esophageal sensitivity, assessed by the multimodal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* HV aged between 18 - 60 years

Exclusion Criteria:

* history of psychiatric disease or a positive first degree psychiatric family history
* pregnancy or lactation
* concomitant administration of any centrally activating medication (anti-depressive medication, hypnotics, sedatives, anxiolytics, …)
* medication affecting esophageal motility
* significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic)
* prior history of esophageal, gastric surgery or endoscopic anti-reflux procedure
* history of gastrointestinal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in sensitivity to thermal stimulation | After 30 minutes after administration buspirone
  To detect changes in thermal stimulation for sensitivity

SECONDARY OUTCOMES:
Change in sensitivity to mechanical stimulation | After 45 minutes after administration buspirone
  To detect changes in mechanical stimulation for sensitivity
Change in sensitivity to electrical stimulation | After 60 minutes after administration buspirone
  To detect changes in electrical stimulation for sensitivity
Change in sensitivity to chemical stimulation | After 75 minutes after administration buspirone
  To detect changes in chemical stimulation for sensitivity
Change in positive and negative affect score | At the beginning of the study and at the end of the multimodal stimulation
  to detect change in affect of the multimodal stimulation
Change in state trait and anxiety score | At the beginning of the study and at the end of the multimodal stimulation
  to detect changes in the score due to the multimodal stimulation

IPD SHARING:
Plan to Share IPD: No